CLINICAL TRIAL: NCT04403035
Title: Comparison of the ID NOW and Accula Point-of-Care Assays for the Detection of Severe Acute Respiratory System CoV-2 (SARS-CoV-2)
Brief Title: Comparison of the ID NOW and Accula Point-of-Care Assays for Detection of COVID-19
Status: Withdrawn | Type: Observational
Why Stopped: Unable to get adequate resources to do the study
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 1599159
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2020-07

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ID NOW vs. Acccula arm: Each patient serves as his or her own control. The ID NOW test is the one that is being currently used (i.e. the control) and the Accula test is the newer test being evaluated.
  Interventions: Diagnostic Test: ID NOW vs. Accula

INTERVENTIONS:
Diagnostic Test: ID NOW vs. Accula — Comparison of the ID Now assay vs. the Accula assay in detecting Covid-19.

SUMMARY:
This study is a comparison of the ID Now COVID-19 (Abbott) assay to the Accula SARS-CoV-2 (Mesa Biotech) assay to assist in the identification of infection with COVID-19. The tests will be compared for sensitivity, specificity, positive predictive value and negative predictive value.

DETAILED DESCRIPTION:
In response to the pandemic, the Food and Drug Administration (FDA) approved several platforms under emergency use authorization (EUA). These platforms do not have full FDA approval and may be used for COVID-19 testing temporarily in a clinical laboratory until the manufacturer receives full FDA clearance for use in the U.S.

Two point of care (POC) platforms with current EUA approval are the ID NOW COVID-19 (Abbott) and the Accula SARS-CoV-2 tests (Mesa Biotech). Both tests are designated as clinical laboratory improvement amendments (CLIA) waived complexity. POCs play a vital role in the diagnosis of COVID-19, especially in laboratories and clinics where testing including molecular assays and serology is not available.

The purpose of this study is to compare SARS-CoV-2 results from clinical specimens on the ID NOW and the Accula systems. If the Accula system is comparable or demonstrates superior test parameters including sensitivity, then this assay may potentially assist in improving turnaround times for COVID-19 results and facilitate reinstating elective procedures.

Patients with orders for rapid Covid-19 testing and who have consented to participate will be included. For these patients one additional clinical specimen, a nasal specimen will be collected from the patient at the same time as the initial specimen for the ID NOW. If there is a discrepancy between the ID NOW and Accula test results, an additional specimen (nasal) will be collected from the patient, if possible (i.e. if the patient remains in-house) to confirm the COVID-19 results. We will also include patients who did not have an initial swab but tested positive by PCR. They will be swabbed by both systems.

This study will evaluate accuracy by comparing Accula results to the ID NOW, precision (reproducibility) by repeating select specimens with different users and on different analyzers, limit of detection by diluting commercial SARS-CoV-2 controls with a known concentration and cross-reactivity by testing known respiratory viruses (including influenza A, B and RSV) on the Accula.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 testing has been ordered in the Emergency Dept. or for inpatients in the hospital or patient has already tested positive via PCR.
* Adult patients
* Consent obtained

Exclusion Criteria:

* Testing not ordered or tested negative via PCR.
* Children
* Do not consent

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with orders for rapid COVID-19 testing who have consented to participate will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-05-09 (Estimated)

PRIMARY OUTCOMES:
Test characteristics | 3 months
  Comparison of accuracy, sensitivity, specificity, and positive and negative predictive values between the two assays.

CONTACTS AND LOCATIONS:
Overall Officials: Melphine Harriott, PhD, Principal Investigator — Ascension St. John Hospital, Detroit, Michigan
Locations (1):
- Ascension St. John Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Accula SARS-CoV-2 Test IFU (EUA). Mesa Biotech, 2020.
- [Result] ID NOW COVID-19 Assay IFU (EUA). Abbott, 2020.
- [Result] Laboratory testing for 2019 novel coronavirus (2019-nCoV) in suspected human cases: Interim guidance. World Health Organization. 19 March 2020.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04403035/Prot_SAP_002.pdf
  • Informed Consent Form (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04403035/ICF_003.pdf